CLINICAL TRIAL: NCT00571077
Title: Electrical Impedance Scanning of Thyroid Nodules Prior to Thyroid Surgery: a Prospective Study
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Aviram Nissan, Hadassah-Hebrew University Medical Center
Other Study IDs: 1-31-7-02; EIS-T-02
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2007-12

CONDITIONS: Thyroid Neoplasms; Thyroid Nodules
Keywords: Thyroid neoplasms; thyroid nodules; electrical impedance scanning
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens are retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: This is a a single arm study evaluating the efficacy and accuracy of EIS in detecting malignant thyroid nodules.
  PAtients with thyroid nodules scheduled for surgery will undergo EIS examination.
  Interventions: Device: Electrical Impedance Scanning (EIS) of the Thyroid gland

INTERVENTIONS:
Device: Electrical Impedance Scanning (EIS) of the Thyroid gland — Patients will be examined in the supine position. A cylinder electrode conveying 2.5V electrical current will be held by the patient. The patient will be scanned by a probe (similar to an ultrasound probe. The examination takes 5 minutes and there is no risk or discomfort.

SUMMARY:
Patients over the age of 18 with thyroid nodules scheduled for surgery will undergo EIS scan. Each node will be scanned and graded form 1-5 (1=benign, 5=malignant). Results will be compared with final histopathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 with thyroid nodules scheduled for surgery.

Exclusion Criteria:

* Pregnant patients
* PAtients with electrical powered devices (cardiac pacemakers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 with thyroid nodules scheduled for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2002-01; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of EIS | 5 years

SECONDARY OUTCOMES:
NPV and PPV of EIS of the thyroid | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aviram Nissan, MD, Principal Investigator — Hadassah Medical Organization; Alexander Stojadinovic, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (2):
- Walter Reed Army MEdicla Center, Washington D.C., District of Columbia, United States
- Hadassah-Hebrew University Medical Center, Jersualem, Israel

REFERENCES:
- [Derived] Nissan A, Peoples GE, Abu-Wasel B, Adair CF, Prus D, Howard RS, Lenington SG, Fields SI, Freund HR, Peretz T, Burch HB, Shriver CD, Stojadinovic A. Prospective trial evaluating electrical impedance scanning of thyroid nodules before thyroidectomy: final results. Ann Surg. 2008 May;247(5):843-53. doi: 10.1097/SLA.0b013e318165c757. PMID 18438123